CLINICAL TRIAL: NCT00216216
Title: Pemetrexed (Alimta) in Patients With Chemosensitive and Chemoresistant Relapsed Small Cell Lung Cancer: A Hoosier Oncology Group Phase II Study (LUN04-78)
Brief Title: Pemetrexed in Patients With Chemosensitive and Chemoresistant Relapsed Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The results from the interim analysis were not favorable to continue this trial.
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Eli Lilly and Company (Industry); Walther Cancer Institute (Other)
Responsible Party: Nasser Hanna, M.D., Hoosier Oncology Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG LUN04-78
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2011-04

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Pemetrexed for patients with chemosensitive and chemoresistant relapsed small cell lung cancer.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed 500 mg/m2 IV q 3 weeks

SUMMARY:
Patients with relapsed or chemotherapy-refractory SCLC have a dismal prognosis. Unfortunately, available treatments result in few durable responses. Pemetrexed is a well-tolerated agent, which is active in NSCLC. Since chemotherapy agents, which are active in NSCLC, are usually also active in SCLC, this trial will examine the efficacy and activity of pemetrexed in this palliative setting

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Pemetrexed 500 mg/m2 i.v. q 3 wks

All patients will also receive folic acid 350-1000 mcg. po once daily beginning approximately 1 week prior to the first dose of pemetrexed and continuing until completion of pemetrexed, Vitamin B12 1000 mcg. IM every 9 weeks beginning approximately 1 week prior to the first dose of pemetrexed and continuing until completion of pemetrexed, and dexamethasone 4 mg po bid the day before, the day of, and the day following each treatment with pemetrexed

Chest x-ray will be performed prior to each cycle (if other disease assessment by imaging is not performed) in order to ensure patients are not rapidly progressing.

Cycles are repeated every 3 weeks for up to 6 cycles or PD or intolerable side effects.

Performance Status: ECOG 0, 1, or 2

Life Expectancy: Not specified

Hematopoietic:

* WBC > 3000/mm3
* ANC > 1500/mm3
* Platelet count > 100,000/mm3
* Hemoglobin > 8 g/dL

Hepatic:

* Bilirubin < 1.0 X upper limit of normal
* Aspartate aminotransferase (AST, SGOT) < 2.5 x upper limit of normal. AST may be < 5 x upper limit of normal for patients with liver metastasis

Renal:

* Creatinine clearance of > 45 ml/ min (by Cockcroft-Gault)

Cardiovascular:

* No unstable or uncompensated cardiovascular conditions

Pulmonary:

* No unstable or uncompensated respiratory conditions

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of neuroendocrine cancers (including small cell cancers of any site [including lung] or poorly differentiated neuroendocrine cancers of the lung with (unidimensionally) measurable disease as per the RECIST criteria
* Chemoresistant or chemosensitive disease
* Patients must have received treatment with at least one but not more than 2 prior chemotherapy regimens, including one regimen containing a platinum agent
* Radiation therapy must have completed their radiation at least 14 days prior to being registered for protocol therapy, and toxicities due to radiation must have recovered to < grade 1 or baseline prior to registration
* Negative pregnancy test

Exclusion Criteria:

* No clinically significant infections as judged by the treating investigator
* No symptomatic CNS metastasis
* No radiation to > 25% of the marrow containing spaces
* No previous treatment with pemetrexed
* No uncontrolled pleural effusions
* No current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2005-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
- To estimate the clinical benefit rate (CR, PR, SD) of pemetrexed in two patient populations with small cell lung cancer: chemosensitive and chemoresistant relapsed independently. | 12 months

SECONDARY OUTCOMES:
To determine the toxicity of pemetrexed; To estimate the time to disease progression; To estimate overall survival | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (16):
- United States (16):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen Health System, Goshen, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Community Regional Cancer Center, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Center for Cancer Care, Inc., P.C., New Albany, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Northern Indiana Oncology Associates, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Cancer Center, Omaha, Nebraska

REFERENCES:
- [Result] Jalal S, Ansari R, Govindan R, Bhatia S, Bruetman D, Fisher W, Masters G, White A, Stover D, Yu M, Hanna N; Hoosier Oncology Group. Pemetrexed in second line and beyond small cell lung cancer: a Hoosier Oncology Group phase II study. J Thorac Oncol. 2009 Jan;4(1):93-6. doi: 10.1097/JTO.0b013e31818de1e6. PMID 19096313
- See also: Hoosier Oncology Group Home Page — http://hoosieroncologygroup.org